CLINICAL TRIAL: NCT06229808
Title: New Design; Investigation of the Effect of Multifunctional Birthing Ball on Perineal and Sacral Pain and Duration of Labor in the First Two Stages of Labor
Brief Title: The Effect of the Multifunctional Birthing Ball on Labor Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Betul Mammadov, Assistant Professor, Near East University, Turkey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: YDU/2021/93-1378
Record Dates: First submitted 2024-01-03; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Labor Pain
Keywords: Labor Pain; Birth Ball; Active Delivery; Massage; Perineal Warming
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multifunctional Birthing Ball group (Experimental): Massages will be applied to the experimental group in the first stage of labor for 30 minutes each at the end of the latent, active and transition phases (cervical dilatation 3-4 cm, 5-7 cm, 8-10 cm), respectively.
  Perineal heating application is planned to be performed at least twice until the delivery occurs as 20 minutes of application and 20 minutes of tissue rest periods when the second stage of labor begins (the duration of this stage may reach 2 hours in primiparous women).
  Interventions: Device: Multifunctional Birthing ball
- Control group (No Intervention): No intervention will be applied

INTERVENTIONS:
Device: Multifunctional Birthing ball — In order to reduce low back pain in labor, massages will be applied to the experimental group in the first stage of labor for 30 minutes each at the end of the latent, active and transition phases (cervical dilatation 3-4 cm, 5-7 cm, 8-10 cm), respectively.
  Perineal heating application is planned to be performed at least twice until the delivery occurs as 20 minutes of application and 20 minutes of tissue rest periods when the second stage of labor begins (the duration of this stage may reach 2 hours in primiparous women).
  Arms: Multifunctional Birthing Ball group

SUMMARY:
Objective: By using the newly designed multifunctional birthing ball, it is aimed to reduce the intense perineal and sacral pain in the first and second stages of labor, to prevent perineal tears, pain and episiotomy opening with perineal heating, to take advantage of the positive effects of the birthing ball on the pelvis to support active labor and shorten the duration of labor, and to increase the satisfaction of mothers with labor by reducing anxiety and pain.

Materials and Methods: The multifunctional birthing ball will support the active movements of the pregnant woman, as well as warming the perineum while providing lumbar and back massage. The multifunctional birthing ball was developed by researchers and manufactured by the Near East University 3D Lab. The bottom of the ball is made of flexible and explosion-proof material filled with air. The purpose of the ball is to enable the pregnant woman to make swinging and bouncing movements during active labor. The massager and heating pad will be controlled by a single electronic circuit. Three different massage modes can be selected: continuous, intermittent and fluctuating. The heating pad can be turned on and off with a single button and the temperature can be adjusted (decrease-increase). To prevent overheating and tissue damage, a maximum temperature of 42 °C was fixed on the control. The inner padding is made of a material that protects both the massager and the heating pad from external factors and also serves as a seat. The shape of the device is designed to ensure that the massager is in full contact with the waist when the pregnant woman sits on the ball. The coating of the massage chair and heating pad is made of cleanable material suitable for hospital use.

DETAILED DESCRIPTION:
This study was designed to experimentally investigate the effect of a multifunctional birthing ball on perineal pain, sacral pain, total duration of labor, perineal tears, and women's satisfaction with the birth experience during the first and second stages of labor in pregnant women who will deliver vaginally. Pregnant women to be included in the experimental and control groups should meet the following criteria:

* First-time mothers
* At term (37-42 weeks of gestation)
* Single fetal gestation
* Cervical dilatation of 3 cm or greater
* Expected spontaneous delivery
* No pregnancy complications or systemic diseases
* No history of cephalopelvic disproportion, placenta previa, placental abruption, or fetal distress
* Willingness to participate in the study
* Age between 18 and 35 years

Experimental Intervention Participants in the experimental group will receive massages using a multifunctional birthing ball during the first stage of labor. Massages will be administered for 30 minutes each at the end of the latent, active, and transition phases (cervical dilatation 3-4 cm, 5-7 cm, and 8-10 cm, respectively). Visual Analog Scale (VAS) scores will be evaluated three times in each phase to assess low back pain. In the control group, VAS scores will be evaluated three times without massage application for the same periods.

Perineal Heating Application

Perineal heating application will be initiated when the second stage of labor begins and will continue until delivery. The heating application will consist of 20 minutes of application followed by 20 minutes of tissue rest. VAS scores will be evaluated two times during these stages to determine perineal pain. In the control group, VAS scores will be evaluated twice without heating application for the same periods.

Postpartum Evaluation

During the postpartum period, each participant will complete a 30-question "Postpartum Interview Form" that will address questions related to the status of perineal integrity at the end of labor, overall childbirth experience, and satisfaction with the birth process. Additionally, each participant will complete the "Birth Satisfaction Scale" - a 30-item questionnaire designed to assess the woman's satisfaction with her birth experience.

ELIGIBILITY:
Inclusion Criteria:

* First-time mothers
* At term (37-42 weeks of gestation)
* Single fetal gestation
* Cervical dilatation of 3 cm or greater
* Expected spontaneous delivery
* No pregnancy complications or systemic diseases
* Age between 18 and 35 years

Exclusion Criteria:

* Non-pregnancy related chronic illness
* Pregnancy-related illness
* Pregnancy complications

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Birth pain is a pain experienced only by women.
Enrollment: 40 (Actual)
Dates: Start 2022-01-02 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Evaluating pain scores by performing lumbar massage with the massage chair on the birthing ball in order to reduce the back pain experienced during birth. | during the intervention
  In order to reduce the back pain experienced during birth, the experimental group received massages in the first stage of birth, respectively; It will be applied for 30 minutes at the end of the latent, active and transition phases (cervical dilatation 3-4 cm, 5-7 cm, 8-10 cm). To determine low back pain at birth, VAS (visual analogue scale) scores will be evaluated a total of three times at all these stages. In the control group, VAS scores will be evaluated three times without massage application for the same period of time.
Evaluating perineal pain with perineal heating application | during the intervention
  Perineal heating application is planned to be performed at least twice when the second phase of labor begins (in primiparas, this phase may last up to 2 hours), with a 20-minute application and a 20-minute tissue rest period until birth. To determine perineal pain, VAS (visual analogue scale) scores will be evaluated twice in all these stages. In the control group, VAS scores will be evaluated twice at the same time without heating.
Applying the "Birth Satisfaction Scale" to measure the woman's satisfaction with her birth experience in the postpartum period. | immediately after the intervention
  Finally, in the postpartum period, the "Birth Satisfaction Scale" consisting of 30 items will be filled in to measure the woman's satisfaction with her birth experience. The original "Birth Satisfaction Scale (BSS)" was developed by Caroline Hollins in 2009. A Turkish validity and reliability study was conducted by Cosar Cetin F. and his colleagues in 2015. Responses to this scale, which is a 5-point Likert type; Absolutely I agree. 5; I agree. 4; I'm undecided 3; Disagree 2; Strongly Disagree: scores as 1. In the scale items; Items 4, 8, 12, 15, 16, 17, 19, 20, 21, 23, 25, and 29 are scored as reversed items. The total number of points to be obtained from the scale varies between 30 and 150 points. Subthemes in the scale were determined as quality of care, birth environment, adequate support and relationships with health professionals. High scores from the scale indicate that the woman is more satisfied with birth.

CONTACTS AND LOCATIONS:
Locations (1):
- Near East University, Nicosia, Cyprus